CLINICAL TRIAL: NCT00142831
Title: Effectiveness of Bupropion Used in Combination With the Nicotine Replacement Patch and Cognitive Behavioral Therapy for Treating Nicotine Dependent Individuals - 1
Brief Title: Bupropion as an Adjunct to the Nicotine Patch Plus CBT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Maurizio Fava, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-11512-1; R01-11512-1; DPMC
Record Dates: First submitted 2005-09-01; First posted 2005-09-02 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2008-08

CONDITIONS: Tobacco Use Disorder
Keywords: nicotine dependence
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Drug Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Bupropion-SR, 150 mg/day x 3 days, then 300 mg/day for 13 weeks
  Interventions: Drug: Pharmacotherapies for Smoking Cessation
- 2 (Placebo Comparator): Identical Placebo
  Interventions: Drug: Pharmacotherapies for Smoking Cessation

INTERVENTIONS:
Drug: Pharmacotherapies for Smoking Cessation — Bupropion-SR or Identical Placebo

SUMMARY:
Existing and new pharmacotherapies along with prevention efforts are key to improving smoking cessation rates and reducing the premature morbidity and mortality associated with tobacco use. A number of individuals suffer from both nicotine dependence and depression. The purpose of this study is to determine the effectiveness of bupropion used in combination with the nicotine replacement patch and cognitive behavior therapy (CBT) in treating nicotine dependent individuals also diagnosed with depression.

DETAILED DESCRIPTION:
Smoking cessation treatment is highly cost effective and pharmacotherapy is universally recommended for treatment of nicotine dependence. However, the majority of smokers are unable to quit even with treatment. Existing and new pharmacotherapies along with prevention efforts are key to improving smoking cessation rates and reducing the premature morbidity and mortality associated with tobacco use. The purpose of this study is to examine the effectiveness of bupropion as an addition to a standard smoking cessation treatment of CBT and nicotine replacement. In addition, this study will determine if bupropion improves an individual's odds of quitting smoking, and whether this is achieved through its impact on negative mood states associated with depression.

Participants in this double-blind study will be randomly assigned to receive either bupropion or placebo. CBT sessions and individual meetings with a study physician will last for 13 weeks. Treatment with either bupropion or placebo will begin at the first CBT meeting and will continue for 13 weeks. Treatment with the nicotine replacement patch will begin at the second CBT meeting and will continue for 10 weeks. Participants will have monthly follow-up visits throughout the year following Week 13. During the follow-up period, participants will continue to take either bupropion or placebo but will no longer undergo CBT or nicotine replacement. If participants are unable to quit smoking, or become more depressed during the follow-up phase, they will be offered treatment with Zoloft, and will continue to be monitored for the duration of the follow-up year. If participants have been unsuccessful in using Zoloft, they will be offered another antidepressant at the judgement of the clinician.

ELIGIBILITY:
Inclusion Criteria:

* Smokes at least 10 cigarettes per day for at least the past 2 years
* Meets DSM-IV criteria for nicotine dependence, as determined by the Fagerstrom Nicotine Tolerance Questionnaire
* Meets DSM-IV diagnoses of unipolar depressive disorders (major depression, dysthymia, and minor depression)

Exclusion Criteria:

* Current suicidal or homicidal risk
* Serious illness, including cardiovascular, liver, kidney, respiratory, endocrine, neurologic, or hematologic disease
* Untreated peptic ulcer
* Life-threatening arrhythmia, cerebrovascular, or cardiovascular event within the 6 months prior to enrollment
* Severe respiratory compromise, as defined as a FEV-1 less than 1.0 L/min and/or pO2 less than 60 or pCO2 less than 45
* Currently using nicotine-containing products (e.g., cigar, pipe, snuff, nicotine gum)
* History of a seizure disorder
* Current DSM-IV diagnosis of organic mental disorder, schizophrenia, delusional disorder, psychotic disorder, bipolar disorder, or antisocial personality disorder
* Current DSM-IV diagnosis of substance abuse or dependence disorders within the year prior to enrollment
* Current eating disorder, including anorexia nervosa and bulimia nervosa
* History of multiple adverse drug reactions or allergy to bupropion
* Mood congruent or mood incongruent psychotic features
* Current use of other psychotropic drugs (with the exception of hypnotics and benzodiazepines at stable doses for at least six months prior to enrollment or current use of nonbenzodiazepine hypnotics such as Ambien and Sonata)
* Clinical or laboratory evidence of hypothyroidism
* Currently seeking treatment for smoking cessation
* History of skin diseases (e.g., psoriasis), skin allergies, or strong reactions to topical preparations, medical dressings, or tapes
* Currently using topical drugs
* Pregnant
* Not using adequate methods of contraception

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 293 (Actual)
Dates: Start 1999-04; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
7 day point prevalence of cigarette abstinence; measured at Week 13 and on a weekly basis | Weekly, and 13 weeks after beginning study medication (Week 13).

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Fava, M.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Hajizadeh A, Howes S, Theodoulou A, Klemperer E, Hartmann-Boyce J, Livingstone-Banks J, Lindson N. Antidepressants for smoking cessation. Cochrane Database Syst Rev. 2023 May 24;5(5):CD000031. doi: 10.1002/14651858.CD000031.pub6. PMID 37230961